CLINICAL TRIAL: NCT01058291
Title: Phase 3 Study of KW-6500 (Placebo-Controlled Double-Blind Crossover Comparative Study in Patients With Parkinson's Disease)
Brief Title: Placebo-Controlled Double-Blind Crossover Comparative Study of KW-6500
Acronym: 6500-004
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6500-004
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- KW-6500 (Experimental)
  Interventions: Drug: KW-6500
- KW-6500 Placebo (Placebo Comparator)
  Interventions: Drug: KW-6500 Placebo

INTERVENTIONS:
Drug: KW-6500 — Twelve weeks subcutaneous injection of 1 to 6 mg for the OFF state
  Other Names: Apomorphine hydroshloride (USAN)
  Arms: KW-6500
Drug: KW-6500 Placebo — Twelve weeks subcutaneous injection for the OFF state
  Arms: KW-6500 Placebo

SUMMARY:
This is a placebo-controlled double-blind crossover comparative study of KW-6500 in Parkinson's disease patients with motor response complications on levodopa therapy. The efficacy of KW-6500 is evaluated using the change of UPDRS part III score at double blind period after 12 weeks subcutaneous self-injections.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given written informed consent
* Patients who have Parkinson's disease
* Patients who have been on a stable regimen of levodopa plus at least one other antiparkinsonian agent and who have OFF state
* Patients who meet stage 4 or 5 while in the OFF state and stage 0 to 3 while in the ON state on the Modified Hoehn and Yahr Scale
* Patients who have experienced a 30% or more improvement in Unified Parkinson's Disease Rating Scale (UPDRS) partⅢ score when tested for responsiveness to levodopa during the baseline period
* Patients who have at least one OFF state per day
* Patients who can understand the expression of OFF state, ON state, and dyskinesia
* Patients or their families have a desire for self-injection of KW-6500

Exclusion Criteria:

* Patients with an illness of the cardiac, hematologic, hepatic, renal, pancreatic, metabolic, respiratory, gastrointestinal, endocrinologic, or neurologic system (excluding Parkinson's disease)
* Patients with orthostatic hypotension
* Patients with a history of intolerance to morphine or its derivatives, sulfur, sulfur-containing pharmaceutical products, or sulfite
* Patients with a history of malignant syndrome
* Patients with a diagnosis of cancer or evidence of continued disease
* Patients who do not test negative in the direct Coombs' test
* Pregnant or lactating women, women who are planning to have children, women who test positive in the pregnancy test, or women who cannot adhere to a reliable method of contraception
* Patients who have received MAO inhibitors except selegiline
* Patients with a history of mental disease (excluding psychiatric symptoms associated with Parkinson's disease)
* Patients with a Mini-Mental State Examination score of 23 or less
* Patients who are taking antipsychotics or central dopamine antagonists (excluding domperidone)
* Patients who are receiving methyldopa or 5-HT3 receptor antagonists
* Patients who are receiving reserpine or papaverine
* Patients who have had a neurosurgical operation for Parkinson's disease
* Patients who have had transcranial magnetic stimulation
* Patients with a history of drug or alcohol abuse or dependence

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The raw score change in UPDRS part III score | At the double blind period

SECONDARY OUTCOMES:
The percent score change in UPDRS part III score and response ratio | At the double blind period

CONTACTS AND LOCATIONS:
Locations (1):
- Ehime University Hospital, Tōon, Ehime, Japan